CLINICAL TRIAL: NCT02192580
Title: Oral Omega-3 for Reduction of Kidney Scar Due to Pyelonephritis in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Azadeh Eshraghi, Clinical Pharmacist, Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Shahid Behesti University
Record Dates: First submitted 2014-07-13; First posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Acute Pyelonephritis(APN)
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 (Active Comparator): omega-3 (DHA+EPA) in divided 3 times/day in addition to standard regimens: Children less than 18 kg:26 mg/kg EPA and 11 mg/kg DHA Children 18-24 kg:504 mg EPA and 216 mg DHA Children 25-32 kg:672 mg EPA and 288 mg DHA Children 33-41 kg:840 mg EPA and 360 mg DHA Children 5-15 years:1000 mg EPA and 878 mg DHA omega-3 in divided 3 times/day in addition to standard regimens
  Interventions: Drug: Omega-3
- Control (No Intervention): control group received just standard regimens without omega-3

INTERVENTIONS:
Drug: Omega-3 — Children less than 18 kg:26 mg/kg EPA and 11 mg/kg DHA Children 18-24 kg:504 mg EPA and 216 mg DHA Children 25-32 kg:672 mg EPA and 288 mg DHA Children 33-41 kg:840 mg EPA and 360 mg DHA Children 5-15 years:1000 mg EPA and 878 mg DHA omega-3 in divided 3 times/day in addition to standard regimens
  Arms: Omega-3

SUMMARY:
Urinary tract infections (UTI) are a common and important clinical problem in childhood.Upper urinary tract infections (ie, acute pyelonephritis) may lead to renal scarring, hypertension, and end-stage renal disease.Pathogenesis of acute pyelonephritis (APN) is associated with urinary tract anatomy and function, bacterial virulence factors, the host innate immune system and production of free radicals. Oxygen-free radicals and oxidative stress play a role in renal scar formation after an APN. Oxygen-free radical scavengers and antioxidants can reduce tissue damage and renal scaring during acute pyelonephritis.we want to publish a study that indicates that antioxidant therapy with omega-3 given to children with pyelonephritis may indeed lower the risk for renal scarring.

Several studies show that omega-3 alleviated oxidative stress and inflammation.This study is a simple randomized clinical trial (RCT) evaluating the effect of omega-3 in addition to antibiotic on preventing renal scaring after acute pyelonephritis in children. This randomized clinical trial on 60 patients in 2 groups (intervention & control) is conducted.Children aged 1 month to 10 years with positive urine culture, clinical findings, and 99mTc-dimercaptosuccinic acid (DMSA) scintigraphy-based evidence in favor of acute pyelonephritis were enrolled into a clinical trial. Patients with neurogenic bladder, systemic hypertension, obstructive uropathy and high grade vesicouretera are excluded.Patients in Intervention group are administered omega-3 based on body weight in divided doses in addition to antibiotic regimens and patients in control group received antibiotic regimens without omega-3. Primary outcome is the development of renal scar by doing DMSA renal scan on the 7th day of admission and four to six months after the intervention and compared between groups.Also,measurement of urinary biomarker of acute kidney injury (NGAL) three days after antibiotic or omega-3 administration for assessing of subsequent scarring in both groups will be done . Secondary outcome is the incidence and severity of renal scarring after pyelonephritis and response to treatment between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month to 10 years with positive urine culture, clinical findings, and 99mTc-dimercaptosuccinic acid (DMSA) scintigraphy-based evidence in favor of acute pyelonephritis

Exclusion Criteria:

* neurogenic bladder,
* systemic hypertension,
* obstructive uropathy,
* High grade vesicoureteral

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Change of 99mTc-dimercaptosuccinic acid (DMSA) scan | Baseline and 4 months

SECONDARY OUTCOMES:
Urinary biomarker of acute kidney injury (NGAL) | 3th day

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Mehrpooya, Ph.D, Principal Investigator — Hamedan University of Medical Sciences; Alaleh Gheisari, Principal Investigator — Pediatric Nephrologist,Isfahan University, Isfahan, Iran; Elham Jafari, Ph.D, Principal Investigator — Isfahan University, Isfahan, Iran; Azadeh Eshraghi, Ph.D, Principal Investigator — Shahid Beheshti University of Medical Sciences; Golnaz Vaseghi, Ph.D, Principal Investigator — Physiology Research Center,Isfahan University of Medical Sciences; Iraj Sedighi, Principal Investigator — Pediatric infectious disease,Hamedan University of Medical Sciences
Locations (1):
- Hamedan University of Medical Sciences, Hamadan, Iran